CLINICAL TRIAL: NCT00622908
Title: A Study to Evaluate the Clinical and Microbial Efficacy of 0.6% ISV-403 Compared to Vehicle in the Treatment of Bacterial Conjunctivitis
Brief Title: Clinical and Microbial Efficacy of ISV403 in Bacterial Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 373
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Results first posted 2009-08-13 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — besifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ISV-403 (Experimental): ISV-403 0.6%
  Interventions: Drug: ISV-403
- Vehicle (Placebo Comparator): Vehicle of ISV-403
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: ISV-403 — 0.6% TID, 5 days
  Other Names: besifloxacin
  Arms: ISV-403
Drug: Vehicle — Vehicle of ISV-403 TID, 5 days
  Arms: Vehicle

SUMMARY:
To evaluate the clinical and microbial efficacy of ISV-403 administered three times a day (TID) for 5 days compared to vehicle three times a day for 5 days in the treatment of bacterial conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Must be at least one year of age.
* Must have signature of subject or legally authorized representative (if subject is under 18 years of age) on the informed Consent Form.
* Must have signature of subject on the Assent Form if subject is 6 to 17 years of age.
* Must have a clinical diagnosis of acute bacterial conjunctivitis and exhibit purulent conjunctival discharge (crusty or sticky eyelids) and redness in at least one eye. A minimum score of 1 should be present for discharge and a minimum score of 1 for either bulbar or palpebral conjunctival injection.
* Must have pinholed visual acuity equal to or better than 20/200 in both eyes. Age appropriate visual acuity testing was to be performed. Every effort was made to obtain a visual acuity measurement in children. If visual acuity was unobtainable in children, it was at the investigator's discretion to meet inclusion criteria.
* Must be willing to discontinue contact lens wear for the duration of the study.
* Must be willing to avoid disallowed medications during the study period.
* Must understand the scope of the study including completion of diary, be willing to follow instructions, and be able to make all required study visits.
* If a subject was a female of childbearing potential, she must utilize reliable contraceptive methods and have a negative pregnancy test.

Exclusion Criteria:

* Any uncontrolled systemic disease or debilitating disease.
* Use of topical ophthalmic solutions including tear substitutes within two hours before and during the study.
* Use of any ophthalmic topical anti-inflammatory agents within 48 hours before and during the study.
* Subjects likely to require antimicrobial therapy with any active respiratory tract infection, urinary tract infection, skin/soft tissue infection, or otitis media.
* Pregnant or nursing females.
* Known hypersensitivity to SS734 or to any of the ingredients in the study medications.
* Known hypersensitivity to fluoroquinolones or to any of the ingredients in the study medications.
* Ocular surgery (including laser surgery) in either eye within the past six weeks.
* Subjects with suspected viral or allergic conjunctivitis (i.e., severe itching or acute follicular conjunctivitis), or any other disease conditions that could interfere with the efficacy and safety evaluations of the study medication.
* Subjects with suspected iritis (i.e., smaller pupil, pain, and photophobia in infected eye).
* History of recurrent corneal erosion syndrome, either idiopathic or secondary to previous corneal trauma or dry eye syndrome.
* Use of any antibiotic within 72 hours of enrollment.
* Any active ulcerative keratitis, specifically any epithelial loss greater than punctate keratitis
* Participation in an ophthalmic drug or device research study within the 30 days prior to entry in this study.
* Subjects who were immune compromised.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2004-12; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Comstock, OD, Study Director — Bausch & Lomb Incorporated

REFERENCES:
- [Derived] DeCory HH, Sanfilippo CM, Proskin HM, Blondeau JM. Characterization of baseline polybacterial versus monobacterial infections in three randomized controlled bacterial conjunctivitis trials and microbial outcomes with besifloxacin ophthalmic suspension 0.6. PLoS One. 2020 Aug 25;15(8):e0237603. doi: 10.1371/journal.pone.0237603. eCollection 2020. PMID 32841261
- [Derived] Comstock TL, Paterno MR, Decory HH, Usner DW. Safety and tolerability of besifloxacin ophthalmic suspension 0.6% in the treatment of bacterial conjunctivitis: data from six clinical and phase I safety studies. Clin Drug Investig. 2010;30(10):675-85. doi: 10.2165/11536720-000000000-00000. PMID 20629472
- [Derived] Karpecki P, Depaolis M, Hunter JA, White EM, Rigel L, Brunner LS, Usner DW, Paterno MR, Comstock TL. Besifloxacin ophthalmic suspension 0.6% in patients with bacterial conjunctivitis: A multicenter, prospective, randomized, double-masked, vehicle-controlled, 5-day efficacy and safety study. Clin Ther. 2009 Mar;31(3):514-26. doi: 10.1016/j.clinthera.2009.03.010. PMID 19393842

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was started on 12/28/04 and last patient last visit was 6/7/05. This study took place at 35 centers in the US.
Pre-assignment Details: 270 subjects were enrolled, 269 were randomized(1 subject refused culture), 118 of which had bacteriologically confirmed acute bacterial conjunctivitis at baseline.
Groups:
- ISV-403: 0.6% ISV-403
Period: Overall Study
Arm/Group | ISV-403 | Vehicle
Started | 137 (Intent to treat population) | 132 (Intent to treat population)
Completed | 134 | 122
Not Completed | 3 | 10
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 1 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Refusal | 0 | 1
Not completed — Termination by study sponser | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ISV-403 | Vehicle | Total
Number analyzed (Participants) | 137 | 132 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (22.3) | 35.1 (22.4) | 34.2 (22.3)
Age, Customized [Number; unit: Participants]
  < 2 years | 2 | 1 | 3
  2 to 19 Years | 44 | 37 | 81
  20 to 59 Years | 71 | 71 | 142
  >/=60 Years | 20 | 23 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 76 | 162
  Male | 51 | 56 | 107
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 116 | 106 | 222
  Asian | 2 | 2 | 4
  Black or African American | 6 | 11 | 17
  Hispanic | 12 | 8 | 20
  Other | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Clinical Resolution of Baseline Bacterial Conjunctivitis (Day 8 or 9)
Description: Resolution of conjunctival discharge, bulbar conjunctival injection and palpebral conjunctival injection.
Time Frame: Visit 3 - day 8 or 9
Population: Intent to treat population, culture confirmed. Missing values and discontinued patients imputed as failures.
Measure: Number; unit: Participants
Arm/Group | ISV-403 | Vehicle
Number analyzed (Participants) | 60 | 56
Participants | 37 | 20

2. Primary Outcome: Eradication of Baseline Pathogens (Day 8 or 9)
Description: Bacterial species eradication of baseline bacterial infection
Time Frame: Visit 3 - Day 8 or day 9
Population: Intent to treat population, culture confirmed. Missing values and discontinued patients imputed as failures.
Measure: Number; unit: Participants
Arm/Group | ISV-403 | Vehicle
Number analyzed (Participants) | 60 | 55
Participants | 54 | 38

3. Secondary Outcome: Clinical Resolution of Baseline Bacterial Conjunctivitis Day 4 (+/- 1 Day)
Description: The absence of conjunctival discharge, bulbar conjunctival injection and palpebral conjunctival injection.
Time Frame: Visit 2 - Day 4 (+/- 1 day)
Population: Intent to treat population, culture confirmed. Missing values and discontinued patients imputed as failures.
Measure: Number; unit: Participants
Arm/Group | ISV-403 | Vehicle
Number analyzed (Participants) | 60 | 56
Participants | 14 | 8

4. Secondary Outcome: Eradication of Baseline Pathogens Day 4 (+/- 1 Day)
Description: Bacterial species eradication of baseline bacterial infection
Time Frame: Visit 2 - Day 4 (+/- 1 day)
Population: Intent to treat population, culture confirmed. Missing values and discontinued patients imputed as failures.
Measure: Number; unit: Participants
Arm/Group | ISV-403 | Vehicle
Number analyzed (Participants) | 60 | 54
Participants | 54 | 28

ADVERSE EVENTS:
Time Frame: Treated period was 5 days
Arm/Group | ISV-403 | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/137 | 1/132
Other Adverse Events (participants affected / at risk) | 45/137 | 46/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISV-403 (N=137) | Vehicle (N=132)
Loss of Consciousness (Nervous system disorders) | 1 (1) | 1 (1) — Dehydration, not related to study medication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISV-403 (N=137) | Vehicle (N=132)
Eye Pain (Eye disorders) | 16 (24) | 8 (24)
Blurred Vision (Eye disorders) | 15 (28) | 13 (28)
Eye Irritation (Eye disorders) | 11 (27) | 16 (27)
Eye Pruritis (Eye disorders) | 3 (12) | 9 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has 45 days to review materials and provide comments back to the investigator.